CLINICAL TRIAL: NCT06105918
Title: Phase 1 Trial to Determine Safety and Feasibility in Treating Biochemical Recurrence Post-Prostatectomy With PSMA PET Guided External Beam Radiotherapy Followed by Consolidative Radioligand Therapy
Brief Title: Radioligand Therapy After PSMA PET Guided External Beam Radiotherapy for Treating Post-Prostatectomy Patients With Biochemically Recurrent Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David M Schuster, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005677; NCI-2023-03480 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00005677 (Other: Emory University Hospital/Winship Cancer Institute); RAD5633-23 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2023-10-10; First posted 2023-10-30 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Prostate Adenocarcinoma
MeSH Terms: interventions — Specimen Handling; Congresses as Topic; Radiation; Lutetium-177; Magnetic Resonance Spectroscopy; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (EBRT, 177Lu-rhPSMA-10.1) (Experimental): Patients undergo EBRT followed by 177Lu-rhPSMA-10.1 IV on study. Patients also receive rhPSMA-7.3 IV with PET/CT at screening and undergo SPECT-CT and collection of blood samples on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Other: Flotufolastat F-18; Drug: Lutetium Lu 177 PSMA-10.1; Procedure: Positron Emission Tomography; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo rhPSMA-7.3 PET/CT and SPECT-CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Other: Flotufolastat F-18 — Given IV
  Other Names: (18F)-rhPSMA-7.3; 18F-rhPSMA-7.3; 18FrhPSMA-7.3; F-18-rhPSMA-7.3; Fluorine F 18 radiohybrid PSMA-7.3; Fluorine F 18 rhPSMA-7.3; Fluorine-18 rhPSMA-7.3; rhPSMA-7.3 (18F)
Drug: Lutetium Lu 177 PSMA-10.1 — Given IV
  Other Names: (177Lu) rhPSMA-10.1; 177Lu Radiohybrid PSMA-10.1; 177Lu rhPSMA-10.1; 177Lu-rhPSMA-10.1
Procedure: Positron Emission Tomography — Undergo rhPSMA-7.3 PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT-CT scan
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This phase I trial tests the safety, side effects and best dose of radioligand therapy (lutetium Lu 177 PSMA-10.1 [177Lu-rhPSMA-10.1]) after prostate specific membrane antigen (PSMA) positron emission tomography (PET)-guided external beam radiotherapy in treating post-prostatectomy patients with prostate cancer that has come back after a period of improvement (recurrent). In this study, radioligand therapy is a radioactive drug called 177Lu-rhPSMA-10.1. It works by binding to PSMA-expressing prostate tumor cells and delivering the radioactive portion of the drug directly to the tumor cells while not harming normal cells. Radiation therapy such as external beam radiotherapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving radioligand therapy with PSMA PET-guided external beam radiotherapy may kill more tumor cells in post-prostatectomy patients with biochemically recurrent prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate the safety and feasibility of treating radiotherapy (RT) prostate cancer patients via addition of lutetium Lu 177 PSMA-10.1 (177Lu-rhPSMA-10.1) in a selected post-prostatectomy population.

II. Analyze dosimetry of radioligand therapy (RLT) after each cycle of 177Lu-rhPSMA-10.1.

EXPLORATORY OBJECTIVE:

I. Determine the feasibility of and develop preliminary data in the correlation of circulating tumor circulating tumor deoxyribonucleic acid (ctDNA) at baseline, after RT, and RLT.

OUTLINE: This is a dose-escalation study of 177Lu-rhPSMA-10.1.

Patients undergo external beam radiation therapy (EBRT) followed by 177Lu-rhPSMA-10.1 intravenously (IV) on study. Patients also receive flotufolastat F-18 (rhPSMA-7.3) IV with positron emission tomography (PET)/computed tomography (CT) at screening and undergo single-photon emission computed tomography (SPECT)-CT and collection of blood samples on study.

Patients follow up 6 weeks after the last 177Lu-rhPSMA-10.1 administration.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate, post radical prostatectomy with detectable prostate specific antigen (PSA)
* Clinical PSMA PET/CT obtained, with findings of pelvic uptake only (prostate bed, pelvic lymph node uptake, or both)
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of 0-2
* Age over 18

Exclusion Criteria:

* Contraindications to radiotherapy (including active inflammatory bowel disease or prior pelvic radiotherapy or prior RLT)
* Risk factors for Lu-rhPSMA radioligand therapy (Baseline >= grade 2 myelosuppression, renal insufficiency [glomerular filtration rate (GFR) < 60 mL/min], or xerostomia)
* Definitive findings of systemic metastasis prior imaging (if obtained) or biopsy (if obtained)
* Unacceptable medical or radiation safety risk
* Unmanageable urinary tract obstruction or hydronephrosis; patients with diagnosed or who are at high risk of urinary retention
* GFR < 60 mL/min or creatinine > 1.5-fold upper limit of normal (ULN)
* Liver enzymes > 5-fold ULN
* Total white cell count less than 2.5 x 10^9 /L
* Platelet count less than 75 x 10^9 /L
* Any baseline grade 2 or above myelosuppression, nephrotoxicity, hepatotoxicity, xerostomia, or gastrointestinal (GI) toxicity
* Severe acute co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization in the last 3 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immunocompromised patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiotherapy and radioligand therapy related adverse events | Up to 6 weeks post last radioligand therapy dose
  Will be summarized descriptively using frequencies and percentages of all captured toxicities by grade and relevance.

SECONDARY OUTCOMES:
Tumor and organ at risk dosimetry | At 1-3 days and 4-7 days post radioligand therapy
  Descriptive statistics will be used to perform the post-hoc dosimetry for tumor as applicable and background organs after each cycle of radioligand therapy.
Circulating tumor deoxyribonucleic acid (ctDNA) differences | Up to 5 years
  Descriptive statistics (number of subject, mean, median, standard deviation, minimum, and maximum) will be used to summarize baseline ctDNA and post-radiotherapy ctDNA. Wilcoxon Signed-Ranks Test or paired samples t-test will be used to perform comparisons.
ctDNA differences | Up to 5 years
  Descriptive statistics (number of subject, mean, median, standard deviation, minimum, and maximum) will be used to summarize post radiotherapy ctDNA and post-radioligand therapy ctDNA. Wilcoxon Signed-Ranks Test or paired samples t-test will be used to perform comparisons.
ctDNA differences | Up to 5 years
  Descriptive statistics (number of subject, mean, median, standard deviation, minimum, and maximum) will be used to summarize baseline ctDNA and post-radioligand therapy ctDNA. Wilcoxon Signed-Ranks Test or paired samples t-test will be used to perform comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: David M Schuster, MD, FACR, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Wurzer A, De Rose F, Fischer S, Schwaiger M, Weber W, Nekolla S, Wester HJ, Eiber M, D'Alessandria C. Preclinical comparison of [177Lu]Lu-rhPSMA-10.1 and [177Lu]Lu-rhPSMA-10.2 for endoradiotherapy of prostate cancer: biodistribution and dosimetry studies. EJNMMI Radiopharm Chem. 2024 Feb 26;9(1):18. doi: 10.1186/s41181-024-00246-2. PMID 38407630